CLINICAL TRIAL: NCT03861884
Title: Cognition and NeuroImaging in neuroDegenerative Disorders (CogNID)
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18NS001
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-02

CONDITIONS: Dementia (Diagnosis)
MeSH Terms: conditions — Dementia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitive assessments: Neurocognitive assessments, Birmingham Cognitive Screen
- MRI at 3T: Brain Imaging: MRI at 3T
  Interventions: Diagnostic Test: Cognitive assessments
- MRI at 7T: Brain imaging: Ultrahigh Field MRI at 7T
  Interventions: Diagnostic Test: Cognitive assessments

INTERVENTIONS:
Diagnostic Test: Cognitive assessments — Cognitive assessment and MRI at 3T and/or 7T
  Other Names: MRI at 3T; MRI at 7T
  Groups: MRI at 3T; MRI at 7T

SUMMARY:
This prospective study aims:

1. to compare cognitive performance in different clinical groups of participants with mild cognitive impairment (MCI) or mild dementia [Alzheimer's Disease (AD), Vascular Cognitive Impairment (VCI) and Fronto-temporal Dementia (FTD)] to determine whether scores reveal differential profiles between the groups,
2. to demonstrate differences in imaging markers between different dementia syndromes and healthy volunteers using ultra high-field MRI at 7T.

DETAILED DESCRIPTION:
The imaging arm of the study include:

1. to demonstrate differences in brain iron levels between different dementia syndromes and healthy volunteers using ultra high-field MRI, quantitative susceptibility mapping (QSM) at 7T.
2. to demonstrate variations in the resting oxygen usage as an important biomarker to discriminate between different dementia syndromes.
3. to demonstrate cerebral blood flow changes in the brain, particularly in the hippocampus region, and its correlation with different dementia syndromes using Arterial Spin Labelling MRI technique.
4. to demonstrate increased blood brain barrier leakage in the brain, particularly in the hippocampus region, and its correlation with Alzheimer's Disease (AD) and Vascular Cognitive Impairment (VCI) using a new dynamic contrast-enhanced MRI (DCE-MRI) technique.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent.
2. Either pathological, genetic or imaging biomarker evidence to suggest Fronto-temporal Lobar Degeneration, Alzheimer's Disease or Vascular Cognitive Impairment, or defined clinical diagnoses.

Exclusion Criteria:

1. Lack of mental capacity to consent to study involvement.
2. Not speaking English before age 5 years.
3. Learning disability.
4. MRI contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer's disease, Frontotemporal dementia, Vascular Cognitive Impairment
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive scales on Birmingham Cognitive Screen (BCoS) Scores | Through study completion (an average of one year)
  cognitive sub scores in relation to clinical phenotype

SECONDARY OUTCOMES:
Structural imaging changes on MRI at 3T | Through study completion (an average of one year)
  Structural volume loss
Susceptibility weighted mapping at 7T | Through study completion (an average of one year)
  Quantitative Susceptibility Mapping

CONTACTS AND LOCATIONS:
Overall Officials: Akram Hosseini, MD, PhD, Principal Investigator — Akram.Hosseini@nuh.nhs.uk
Locations (2):
- United Kingdom (2):
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, Easat Midland
  - Nottingham University Hospitals NHS Trust, Nottingham, East Midland